CLINICAL TRIAL: NCT01140659
Title: Objective Evaluation of Patients With Palmar Hyperhidrosis Submitted to Two Levels of Sympathectomy: T3 and T4.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Augusto Ishy / Thoracic surgeon in the thoracic surgery department of the "Hospital das Clínicas de São Paulo", Faculty of Medicine - University of São Paulo (FMUSP)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 005/05
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-05

CONDITIONS: Hyperhidrosis; Quality of Life
Keywords: Hyperhidrosis; Thoracic sympathectomy; Objective measurement of sweat
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Objective measurement of sweat (Other): We selected 40 patients from February 2007 to May 2009. All participants were randomized into two groups of 20 patients (G3 and G4) and underwent the sympathectomy, being followed for 12 months. We used an objective method for measuring sweat, checking the "TEWL (transepidermal water loss) measured by the "VapoMeter", and evaluated the quality of life before and after the operation. Also studied were: incidence and intensity of the compensatory hyperhidrosis.
  Interventions: Procedure: Video-assisted sympathectomy

INTERVENTIONS:
Procedure: Video-assisted sympathectomy — All participants were randomized into two groups of 20 patients (G3 and G4) and underwent video-assisted sympathectomy, being followed for 12 months. During this period, the subjects completed a questionnaire about quality of life and carried out the measurements of sweat by VapoMeter.
  Other Names: Thoracic sympathectomy; Endoscopic thoracic sympathectomy

SUMMARY:
Compare the results obtained with video-assisted sympathectomy performed in two distinct levels ganglionic (third versus fourth thoracic ganglion) for the treatment of palmar hyperhidrosis, through a blind randomized clinical trial using an objective method to measure the sweat before and after the operation.

DETAILED DESCRIPTION:
Currently, the treatment of choice for treating palmar hyperhidrosis (PH) is video-assisted thoracic sympathectomy (VATS) . This minimally invasive technique has been well standardized and provides adequate results with low morbidity.

The main side effect of VATS is compensatory hyperhidrosis (CH). This is present in most cases and is considered the greatest cause of dissatisfaction. To reduce the risk of CH, various studies have been conducted to compare different levels of ganglion resection. These studies have been based on subjective quantification of sweating (assessment of sweating reported by patients) and on the application of quality-of-life questionnaires.

Recently, tests for the objective evaluation of sweating have been developed to quantify sweating among patients with various diseases, including PH. So far, there have not been any studies comparing the long-term results of thoracic sympathectomy on the third ganglion (G3) versus the fourth ganglion (G4)with objective evaluation to quantify sweating.

The present study was prospective, randomized and blinded, with the objective of comparing the results from VATS at two different resection levels: G3 versus G4. All the patients were followed over a one-year period, and their palmar sweating was quantified using a portable device (VapoMeter) to measure transepidermal water loss (TEWL). In addition, CH was evaluated by applying a specific quality-of-life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being determined to accomplish the procedure, because such a statement depends on the level of discomfort suffered by the patient.
* Absence of previous thoracic surgery.
* Concordance with the completion of informed consent.
* Preoperative normal, including chest radiograph, electrocardiogram, blood count, sodium, potassium, urea, creatinine, glucose and thyroid hormones.

Exclusion Criteria:

* Patients with BMI> 25.
* Pregnancy.
* Younger than 15 and more than 45 years.
* Heart disease that may contraindicate the procedure (congestive heart failure, coronary insufficiency, cardiac arrhythmias, symptomatic, acute myocardial infarction, etc.).
* Acute infections or chronic.
* Bleeding disorder.
* Neoplasms.
* Inflammatory diseases of pulmonary or pleural.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Objective measurement of sweat before and after surgery (video-assisted thoracic sympathectomy) T3 and T4. | 12 months
  We used an objective method for measuring sweat, checking the "TEWL (transepidermal water loss) measured by the"VapoMeter". This is a portable instrument that functions noninvasively. It has a closed measurement chamber that eliminates external interference from air currents and enables precise metering of transepidermal water loss (TEWL). The evaporation rate is calculated from the rise in relative air humidity inside the closed chamber of the device, and this value is quantified in g/m²/h (increase in the water mass per unit time per unit of evaporation area).

SECONDARY OUTCOMES:
Assessment of quality of life. | 12 months
  We evaluated the quality of life before and after operation by questionnaire supplied to patients.
  Quality of life before the treatment was classified into five different levels and calculated as the summed total score from the protocol (range from 20 to 100). When the total was greater than 84, the QOL was considered very poor; from 68 to 83 was considered poor; from 52 to 67 was good; from 36 to 51 was very good; and from 20 to 35 was excellent.
  After the treatment, the patients were asked to grade the improvement in each item of the same QOL questionnaire.
Incidence of the compensatory hyperhidrosis | 12 months
  The incidence of compensatory sweating was reported spontaneously by patients during the postoperative evaluation (1 week, 1 month, 6 months and 12th month).
Intensity of the compensatory hyperhidrosis | 12 months
  The intensity of compensatory hyperhidrosis (CH) reported spontaneously by patients was graded as severe or non-severe. CH was considered severe when the sweat was visible, thereby causing embarrassment and leading to the need to change clothes every day

CONTACTS AND LOCATIONS:
Overall Officials: José Ribas M de Campos, Study Director — Professor of Thoracic Surgery - University of São Paulo - Medical College
Locations (1):
- Faculty of Medicine - University of São Paulo., São Paulo, São Paulo, Brazil